CLINICAL TRIAL: NCT01187433
Title: Immunogenicity and Safety of CYD Dengue Vaccine in Healthy Children and Adolescents Aged 9 to 16 Years in South America
Brief Title: Study of CYD Dengue Vaccine in Healthy Children and Adolescents in South America
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CYD30; UTN: U1111-1111-6073 (Other: WHO)
Record Dates: First submitted 2010-08-20; First posted 2010-08-24 (Estimated); Results first posted 2016-11-11 (Estimated); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Dengue; Dengue Hemorrhagic Fever
Keywords: Dengue; Dengue hemorrhagic fever; CYD Dengue Vaccines
MeSH Terms: conditions — Dengue; Severe Dengue | interventions — Sodium Chloride; Tetanus Toxoid; adacel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dengue Vaccine Group (Experimental): Participants will receive Live, attenuated, recombinant dengue serotype 1 , 2, 3 , and 4 virus vaccine
  Interventions: Biological: Live, attenuated, recombinant dengue serotype 1 , 2, 3 , and 4 virus
- Control Group (Placebo Comparator): Participants will receive a placebo, NaCl 0.9%.
  Interventions: Biological: NaCl 0.9%; Biological: Tetanus toxoid, reduced diphtheria toxoid, acellular pertussis vaccine adsorbed; Biological: Meningococcal A+C vaccine

INTERVENTIONS:
Biological: Live, attenuated, recombinant dengue serotype 1 , 2, 3 , and 4 virus — 0.5 mL, Subcutaneous (SC)
  Other Names: CYD Dengue Vaccine
  Arms: Dengue Vaccine Group
Biological: NaCl 0.9% — 0.5 mL, Subcutaneous
  Arms: Control Group
Biological: Tetanus toxoid, reduced diphtheria toxoid, acellular pertussis vaccine adsorbed — 0.5 mL, Intramuscular
  Other Names: ADACEL®
  Arms: Control Group
Biological: Meningococcal A+C vaccine — 0.5 mL, Intramuscular
  Arms: Control Group

SUMMARY:
The purpose of this study is to generate immunogenicity and safety data in preparation for efficacy studies in Latin America.

Primary Objectives:

* To describe the immune response to dengue viruses before and after each vaccination with CYD dengue vaccine.
* To evaluate the safety of each vaccination with CYD dengue vaccine.

DETAILED DESCRIPTION:
Participants in the Dengue Vaccine Group will receive 3 vaccinations with CYD Dengue vaccine. Participants in the Control Group will receive placebo vaccinations for the first 2 vaccinations, followed by tetanus toxoid, reduced diphtheria toxoid, and acellular pertussis vaccine adsorbed (ADACEL®) (in Venezuela) or Meningococcal A+C vaccine (in Brazil) as a way of providing therapeutic benefit to the participants in the control group.

ELIGIBILITY:
Inclusion Criteria :

* Aged 9 to 16 years on the day of inclusion
* Participant in good health, based on medical history and physical examination
* Provision of assent form/informed consent form signed by the participant and by the parent(s) or another legally acceptable representative
* Participant and parent(s)/legally acceptable representative(s) able to attend all scheduled visits and to comply with all trial procedures
* For a female participant of child-bearing potential, avoid becoming pregnant (use of an effective method of contraception or abstinence) for at least 4 weeks prior to first vaccination until at least 4 weeks after the last vaccination

Exclusion Criteria :

* Personal or family history of thymic pathology (thymoma), thymectomy, or myasthenia
* For a female participant of child-bearing potential, known pregnancy or positive urine pregnancy test at Visit 1
* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding the first trial vaccination
* Breast-feeding woman
* Planned participation in another clinical trial during the present trial period
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroids therapy
* Known systemic hypersensitivity to any of the components of any of the trial vaccines or history of a life-threatening reaction to any of the trial vaccines or to a vaccine containing any of the same substances
* Chronic illness at a stage that could interfere with trial conduct or completion, in the opinion of the Investigator
* Current alcohol abuse or drug addiction that may interfere with the participant's ability to comply with trial procedures
* Receipt of blood or blood-derived products in the preceding 3 months that might interfere with the assessment of immune response
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination
* Planned receipt of any vaccine in the 4 weeks following the first trial vaccination
* Participant deprived of freedom by administrative or court order, or in an emergency setting, or hospitalized without his/her consent
* Febrile illness (temperature ≥ 38.0 ºC) or moderate or severe acute illness/infection on the day of vaccination, according to Investigator judgment
* Thrombocytopenia, bleeding disorder or anticoagulants in the 3 weeks preceding inclusion contraindicating intramuscular vaccination
* Severe diseases with or without fever, convulsions or neurological abnormalities without treatment or in progression.

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2010-08; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (1):
- Vitória, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Result] Dayan GH, Garbes P, Noriega F, Izoton de Sadovsky AD, Rodrigues PM, Giuberti C, Dietze R. Immunogenicity and safety of a recombinant tetravalent dengue vaccine in children and adolescents ages 9-16 years in Brazil. Am J Trop Med Hyg. 2013 Dec;89(6):1058-1065. doi: 10.4269/ajtmh.13-0304. Epub 2013 Nov 4. PMID 24189367
- [Derived] Coronel D, Garcia-Rivera EJ, Rivera DM, Arredondo-Garcia JL, Dietze R, Perroud AP, Cortes M, Bonaparte M, Wang H, Pagnon A, Jantet-Blaudez F, Penalosa LAR, Dayan G, Zambrano B, DiazGranados CA, Noriega F. Immune Response Persistence and Safety of a Booster Dose of the Tetravalent Dengue Vaccine in Adolescents and Adults Who Previously Completed the 3-dose Schedule 4-5 Years Earlier in Latin America: A Randomized Placebo-controlled Trial. Pediatr Infect Dis J. 2020 Oct;39(10):961-968. doi: 10.1097/INF.0000000000002830. PMID 32932330
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 20 August 2010 to 8 December 2011 at 1 clinical site in Brazil.
Pre-assignment Details: A total of 150 participants who met all of the inclusion criteria and none of the exclusion criteria were enrolled and randomized.
Groups:
- CYD Dengue Vaccine Group: Participants received 3 injections of the CYD dengue vaccine, 1 injection each at 0, 6, and 12 months.
- Control Group: Participants received 3 injections of placebo, 1 injection each at 0, 6, and 12 months.
Period: Overall Study
Arm/Group | CYD Dengue Vaccine Group | Control Group
Started | 100 | 50
Completed | 89 | 46
Not Completed | 11 | 4
Not completed — Protocol Violation | 6 | 2
Not completed — Withdrawal by Subject | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CYD Dengue Vaccine Group | Control Group | Total
Number analyzed (Participants) | 100 | 50 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 100 | 50 | 150
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Age Continuous | 12.7 (2.1) | 12.7 (2.2) | 12.7 (2.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 23 | 82
  Male | 41 | 27 | 68
Region of Enrollment [Number; unit: Participants]
  Brazil | 100 | 50 | 150

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Seropositivity Against Each Serotype With the Parental Dengue Virus Strains Before and After Vaccinations With Either CYD Dengue Vaccine or a Placebo
Description: Seropositivity was defined as participants achieving neutralizing antibody titers ≥10 (1/dil) against each serotype and was assessed using the Dengue Plaque Reduction Neutralization Test (PRNT).
Time Frame: Before and 28 days after each injection
Population: Seropositivity was assessed in the Full Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 99 | 49
Percentage of participants
  Serotype 1; Pre-Injection 1 (n=99, 49) | 59.6 | 63.3
  Serotype 1; Post-Injection 1 (n=99, 49) | 79.8 | 69.4
  Serotype 1; Pre-Injection 2 (n=94, 47) | 80.9 | 72.3
  Serotype 1; Post Injection 2 (n=94, 47) | 95.7 | 72.3
  Serotype 1; Pre-Injection 3 (n=90, 46) | 78.9 | 69.6
  Serotype 1; Post-Injection 3 (n=89, 46) | 96.6 | 69.6
  Serotype 2; Pre-Injection 1 (n=99, 49) | 65.7 | 67.3
  Serotype 2; Post-Injection 1 (n=99, 49) | 80.8 | 67.3
  Serotype 2; Pre-Injection 2 (n=94, 47) | 80.9 | 74.5
  Serotype 2; Post-Injection 2 (n=94, 47) | 98.9 | 72.3
  Serotype 2; Pre-Injection 3 (n=90, 46) | 85.6 | 76.1
  Serotype 2; Post-Injection 3 (n=89, 46) | 98.9 | 76.1
  Serotype 3; Pre-Injection 1 (n=99, 49) | 62.6 | 65.3
  Serotype 3; Post-Injection 1 (n=99, 49) | 92.9 | 67.3
  Serotype 3; Pre-Injection 2 (n=94, 47) | 89.4 | 72.3
  Serotype 3; Post-Injection 2 (n=94, 47) | 100.0 | 72.3
  Serotype 3; Pre-Injection 3 (n=89, 46) | 94.4 | 71.7
  Serotype 3; Post-Injection 3 (n=89, 46) | 100.0 | 73.9
  Serotype 4; Pre-Injection 1 (n=99, 49) | 47.5 | 51
  Serotype 4; Post -njection 1 (n=99, 48) | 89.9 | 58.3
  Serotype 4; Pre-Injection 2 (n=94, 47) | 92.6 | 57.4
  Serotype 4; Post-Injection 2 (n=94, 47) | 100.0 | 59.6
  Serotype 4; Pre-Injection 3 (n=88, 46) | 97.7 | 69.6
  Serotype 4; Post-Injection 3 (n=89, 46) | 100.0 | 73.9

2. Primary Outcome: Percentage of Flavivirus Immune Participants With Seropositivity Against Each Serotype With the Parental Dengue Virus Strains Before and After Vaccinations With Either CYD Dengue Vaccine or a Placebo
Description: Seropositivity was defined as participants achieving neutralizing antibody titers ≥10 (1/dil) against each serotype and was assessed using the Dengue Plaque Reduction Neutralization Test (PRNT). Flavivirus immune subjects at baseline are defined as those subjects with ≥10 (1/dil) for at least 1 serotype with the parental dengue virus strain or for the yellow fever titer.
Time Frame: Before and 28 days after each injection
Population: Seropositivity was assessed in the Full Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 80 | 41
Percentage of participants
  Serotype 1; Pre-Injection 1 (n=80, 41) | 73.8 | 75.6
  Serotype 1; Post-Injection 1 (n=80, 41) | 88.8 | 82.9
  Serotype 1; Pre-Injection 2 (n=78, 39) | 91.0 | 87.2
  Serotype 1; Post-Injection 2 (n=78, 39) | 100.0 | 87.2
  Serotype 1; Pre-Injection 3 (n=74, 38) | 87.8 | 81.6
  Serotype 1; Post-Injection 3 (n=73, 38) | 98.6 | 81.6
  Serotype 2; Pre-Injection 1 (n=80, 41) | 81.3 | 80.5
  Serotype 2; Post-Injection 1 (n=80, 41) | 93.8 | 80.5
  Serotype 2; Pre-Injection 2 (n=78, 39) | 92.3 | 89.7
  Serotype 2; Post-Injection 2 (n=78, 39) | 100.0 | 87.2
  Serotype 2; Pre-Injection 3 (n=74, 38) | 91.9 | 89.5
  Serotype 2; Post-Injection 3 (n=73, 38) | 100.0 | 89.5
  Serotype 3; Pre-Injection 1 (n=80, 41) | 77.5 | 78
  Serotype 3; Post-Injection 1 (n=80, 41) | 95.0 | 80.5
  Serotype 3; Pre-Injection 2 (n=78, 39) | 93.6 | 87.2
  Serotype 3; Post-Injection 2 (n=78, 39) | 100.0 | 87.2
  Serotype 3; Pre-Injection 3 (n=74, 38) | 97.3 | 84.2
  Serotype 3; Post-Injection 3 (n=73, 38) | 100.0 | 86.8
  Serotype 4; Pre-Injection 1 (n=80, 41) | 58.8 | 61
  Serotype 4; Post-Injection 1 (n=80, 40) | 95.0 | 70
  Serotype 4; Pre-Injection 2 (n=78, 39) | 94.9 | 69.2
  Serotype 4; Post-Injection 2 (n=78, 39) | 100.0 | 71.8
  Serotype 4; Pre-Injection 3 (n=73, 38) | 98.6 | 81.6
  Serotype 4; Post-Injection 3 (n=73, 38) | 100.0 | 84.2

3. Primary Outcome: Percentage of Flavivirus Naïve Subjects With Seropositivity Against Each Serotype With the Parental Dengue Virus Strains Before and After Vaccinations With Either CYD Dengue Vaccine or a Placebo
Description: Seropositivity was defined as participants achieving neutralizing antibody titers ≥10 (1/dil) against each serotype and was assessed using the Dengue Plaque Reduction Neutralization Test (PRNT). Flavivirus naïve subjects at baseline are defined as those subjects with <10 (1/dil) for all serotypes with parental dengue virus strains and for yellow fever titer.
Time Frame: Before and 28 Days after each injection
Population: Seropositivity was assessed in the Full Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 19 | 8
Percentage of participants
  Serotype 1; Pre-Injection 1 (n=19, 8) | 0.0 | 0
  Serotype 1; Post-Injection 1 (n=19, 8) | 42.1 | 0
  Serotype 1; Pre-Injection 2 (n=16, 8) | 31.3 | 0
  Serotype 1; Post-Injection 2 (n=16, 8) | 75.0 | 0
  Serotype 1; Pre-Injection 3 (n=16, 8) | 37.5 | 12.5
  Serotype 1; Post-Injection 3 (n=16, 8) | 87.5 | 12.5
  Serotype 2; Pre-Injection 1 (n=19, 8) | 0.0 | 0
  Serotype 2; Post-Injection 1 (n=19, 8) | 26.3 | 0
  Serotype 2; Pre-Injection 2 (n=16, 8) | 25.0 | 0
  Serotype 2; Post-Injection 2 (n=16, 8) | 93.8 | 0
  Serotype 2; Pre-Injection 3 (n=16, 8) | 56.3 | 12.5
  Serotype 2; Post-Injection 3 (n=16, 8) | 93.8 | 12.5
  Serotype 3; Pre-Injection 1 (n=19, 8) | 0.0 | 0
  Serotype 3; Post-Injection 1 (n=19, 8) | 84.2 | 0
  Serotype 3; Pre-Injection 2 (n=16, 8) | 68.8 | 0
  Serotype 3; Post-Injection 2 (n=16, 8) | 100.0 | 0
  Serotype 3; Pre-Injection 3 (n=15, 8) | 80.0 | 12.5
  Serotype 3; Post-Injection 3 (n=16, 8) | 100.0 | 12.5
  Serotype 4; Pre-Injection 1 (n=19, 8) | 0.0 | 0
  Serotype 4; Post-Injection 1 (n=19, 8) | 68.4 | 0
  Serotype 4; Pre-Injection 2 (n=16, 8) | 81.3 | 0
  Serotype 4; Post-Injection 2 (n=16, 8) | 100.0 | 0
  Serotype 4; Pre-Injection 3 (n=15, 8) | 93.3 | 12.5
  Serotype 4; Post-Injection 3 (n=16, 8) | 100.0 | 25

4. Primary Outcome: Percentage of Subjects With Seropositivity Against At Least 1, 2, 3, or 4 Parental Dengue Virus Serotypes Before and After Vaccinations With Either CYD Dengue Vaccine or a Placebo
Description: as for outcome 1
Time Frame: Before and 28 days after each injection
Population: Seropositivity was assessed in the Full Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 99 | 49
Percentage of participants
  At least 1 serotype; Pre-Injection 1 (n=99, 49) | 68.7 | 71.4
  At least 1 serotype; Post-Injection 1 (n=99, 49) | 97.0 | 71.4
  At least 1 serotype; Pre-Injection 2 (n=94, 47) | 94.7 | 74.5
  At least 1 serotype; Post-Injection 2 (n=94, 47) | 100.0 | 74.5
  At least 1 serotype; Pre-Injection 3 (n=90, 46) | 98.9 | 78.3
  At least 1 serotype; Post-Injection 3 (n=89, 46) | 100.0 | 78.3
  At least 2 serotypes; Pre-Injection 1 (n=99, 49) | 62.6 | 67.3
  At least 2 serotypes; Post-Injection 1 (n=99, 49) | 91.9 | 71.4
  At least 2 serotypes; Pre-Injection 2 (n=94, 47) | 92.6 | 74.5
  At least 2 serotypes; Post-Injection 2 (n=94, 47) | 100.0 | 72.3
  At least 2 serotypes; Pre-Injection 3 (n=90, 46) | 91.1 | 73.9
  At least 2 serotypes; Post-Injection 3 (n=89, 46) | 100.0 | 76.1
  At least 3 serotypes; Pre-Injection 1 (n=99, 49) | 56.6 | 61.2
  At least 3 serotypes; Post-Injection 1 (n=99, 49) | 81.8 | 65.3
  At least 3 serotypes; Pre-Injection 2 (n=94, 47) | 81.9 | 72.3
  At least 3 serotypes; Post-Injection 2 (n=94, 47) | 98.9 | 70.2
  At least 3 serotypes; Pre-Injection 3 (n=90, 46) | 86.7 | 71.7
  At least 3 serotypes; Post-Injection 3 (n=89, 46) | 98.9 | 71.7
  All 4 serotypes; Pre-Injection 1 (n=99, 49) | 47.5 | 46.9
  All 4 serotypes; Post-Injection 1 (n=99, 49) | 72.7 | 53.1
  All 4 serotypes; Pre-Injection 2 (n=94, 47) | 74.5 | 55.3
  All 4 serotypes; Post-Injection 2 (n=94, 47) | 95.7 | 59.6
  All 4 serotypes; Pre-Injection 3 (n=90, 46) | 76.7 | 63
  All 4 serotypes; Post-Injection 3 (n=89, 46) | 96.6 | 67.4

5. Primary Outcome: Percentage of Flavivirus Immune Subjects With Seropositivity Against At Least 1, 2, 3, or 4 Parental Dengue Virus Serotypes Before and After Vaccinations With Either CYD Dengue Vaccine or a Placebo
Description: as for outcome 2
Time Frame: Before and 28 days after each injection
Population: Seropositivity was assessed in the Full Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 80 | 41
Percentage of participants
  At least 1 serotype; Pre-Injection 1 (n=80, 41) | 85.0 | 85.4
  At least 1 serotype; Post-Injection 1 (n=80, 41) | 97.5 | 85.4
  At least 1 serotype; Pre-Injection 2 (n=78, 39) | 97.4 | 89.7
  At least 1 serotype; Post-Injection 2 (n=78, 39) | 100.0 | 89.7
  At least 1 serotype; Pre-Injection 3 (n=74, 38) | 100.0 | 92.1
  At least 1 serotype; Post-Injection 3 (n=73, 38) | 100.0 | 89.5
  At least 2 serotypes; Pre-Injection 1 (n=80, 41) | 77.5 | 80.5
  At least 2 serotypes; Post-Injection 1 (n=80, 41) | 95.0 | 85.4
  At least 2 serotypes; Pre-Injection 2 (n=78, 39) | 97.4 | 89.7
  At least 2 serotypes; Post-Injection 2 (n=78, 39) | 100.0 | 87.2
  At least 2 serotypes; Pre-Injection 3 (n=74, 38) | 95.9 | 86.8
  At least 2 serotypes; Post-Injection 3 (n=73, 38) | 100.0 | 89.5
  At least 3 serotypes; Pre-Injection 1 (n=80, 41) | 70.0 | 73.2
  At least 3 serotypes; Post-Injection 1 (n=80, 41) | 92.5 | 78
  At least 3 serotypes; Pre-Injection 2 (n=78, 39) | 91.0 | 87.2
  At least 3 serotypes; Post-Injection 2 (n=78, 39) | 100.0 | 84.6
  At least 3 serotypes; Pre-Injection 3 (n=74, 38) | 93.2 | 84.2
  At least 3 serotypes; Post-Injection 3 (n=73, 38) | 100.0 | 84.2
  All 4 serotypes; Pre-Injection 1 (n=80, 41) | 58.8 | 56.1
  All 4 serotypes; Post-Injection 1 (n=80, 41) | 87.5 | 63.4
  All 4 serotypes; Pre-Injection 2 (n=78, 39) | 85.9 | 66.7
  All 4 serotypes; Post-Injection 2 (n=78, 39) | 100.0 | 71.8
  All 4 serotypes; Pre-Injection 3 (n=74, 38) | 85.1 | 73.7
  All 4 serotypes; Post-Injection 3 (n=73, 38) | 98.6 | 78.9

6. Primary Outcome: Percentage of Flavivirus Naïve Subjects With Seropositivity Against At Least 1, 2, 3, or 4 Parental Dengue Virus Serotypes Before and After Vaccinations With Either CYD Dengue Vaccine or a Placebo
Description: as for outcome 3
Time Frame: Before and 28 days after each injection
Population: Seropositivity was assessed in the Full Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 19 | 8
Percentage of participants
  At least 1 serotype; Pre-Injection 1 (n=19, 8) | 0.0 | 0
  At least 1 serotype; Post-Injection 1 (n=19, 8) | 94.7 | 0
  At least 1 serotype; Pre-Injection 2 (n=16, 8) | 81.3 | 0
  At least 1 serotype; Post-Injection 2 (n=16, 8) | 100.0 | 0
  At least 1 serotype; Pre-Injection 3 (n=16, 8) | 93.8 | 12.5
  At least 1 serotype; Post-Injection 3 (n=16, 8) | 100.0 | 25
  At least 2 serotypes; Pre-Injection 1 (n=19, 8) | 0.0 | 0
  At least 2 serotypes; Post-Injection 1 (n=19, 8) | 78.9 | 0
  At least 2 serotypes; Pre-Injection 2 (n=16, 8) | 68.8 | 0
  At least 2 serotypes; Post-Injection 2 (n=16, 8) | 100.0 | 0
  At least 2 serotypes; Pre-Injection 3 (n=16, 8) | 68.8 | 12.5
  At least 2 serotypes; Post-Injection 3 (n=16, 8) | 100.0 | 12.5
  At least 3 serotypes; Pre-Injection 1 (n=19, 8) | 0.0 | 0
  At least 3 serotypes; Post-Injection 1 (n=19, 8) | 36.8 | 0
  At least 3 serotypes; Pre-Injection 2 (n=16, 8) | 37.5 | 0
  At least 3 serotypes; Post-Injection 2 (n=16, 8) | 93.8 | 0
  At least 3 serotypes; Pre-Injection 3 (n=16, 8) | 56.3 | 12.5
  At least 3 serotypes; Post-Injection 3 (n=16, 8) | 93.8 | 12.5
  All 4 serotypes; Pre-Injection 1 (n=19, 8) | 0.0 | 0
  All 4 serotypes; Post-Injection 1 (n=19, 8) | 10.5 | 0
  All 4 serotypes; Pre-Injection 2 (n=16, 8) | 18.8 | 0
  All 4 serotypes; Post-Injection 2 (n=16, 8) | 75.0 | 0
  All 4 serotypes; Pre-Injection 3 (n=16, 8) | 37.5 | 12.5
  All 4 serotypes; Post-Injection 3 (n=16, 8) | 87.5 | 12.5

7. Primary Outcome: Geometric Mean Titer Ratios (GMTRs) Against Each Serotype With the Parental of Dengue Virus Strains Before and After Vaccinations With Either CYD Dengue Vaccine or a Placebo
Description: Geometric mean titer ratios were assessed using the Dengue Plaque Reduction Neutralization Test (PRNT).
Time Frame: Before and 28 days after each injection
Population: Geometric mean titer ratios were assessed in the Full Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer ratio
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 99 | 49
Titer ratio
  Serotype 1; Post-Inj. 1 / Pre-Inj. 1 (n=99, 49) | 4.67 [3.37 to 6.47] | 0.834 [0.699 to 0.994]
  Serotype 1; Post-Inj. 2 / Pre-Inj. 1 (n=94, 47) | 7.26 [5.51 to 9.57] | 2.11 [1.12 to 4]
  Serotype 1; Post-Inj. 2 / Pre-Inj. 2 (n=94, 47) | 1.66 [1.31 to 2.10] | 1.25 [0.801 to 1.94]
  Serotype 1; Post-Inj. 3 / Pre-Inj. 1 (n=89, 46) | 4.92 [3.71 to 6.52] | 1.36 [0.797 to 2.31]
  Serotype 1; Post-Inj. 3 / Pre-Inj. 2 (n=89, 46) | 1.07 [0.828 to 1.39] | 0.793 [0.508 to 1.24]
  Serotype 1; Post -nj. 3 / Pre-Inj. 3 (n=89, 46) | 1.48 [1.25 to 1.74] | 0.706 [0.607 to 0.821]
  Serotype 2; Post-Inj. 1 / Pre-Inj. 1 (n=99, 49) | 4.15 [3.07 to 5.59] | 0.733 [0.639 to 0.84]
  Serotype 2; Post-Inj. 2 / Pre-Inj. 1 (n=94, 47) | 6.80 [5.46 to 8.45] | 1.75 [0.956 to 3.21]
  Serotype 2; Post-Inj. 2 / Pre-Inj. 2 (n=94, 47) | 1.97 [1.56 to 2.50] | 0.981 [0.66 to 1.46]
  Serotype 2; Post-Inj. 3 / Pre-Inj. 1 (n=89, 46) | 6.21 [4.96 to 7.78] | 1.68 [1.06 to 2.66]
  Serotype 2; Post-Inj. 3 / Pre-Inj. 2 (n=89, 46) | 1.78 [1.39 to 2.28] | 0.944 [0.646 to 1.38]
  Serotype 2; Post-Inj. 3 / Pre-Inj. 3 (n=89, 46) | 1.40 [1.16 to 1.69] | 0.851 [0.734 to 0.986]
  Serotype 3; Post-Inj. 1 / Pre-Inj. 1 (n=99, 49) | 6.50 [5.01 to 8.45] | 0.916 [0.673 to 1.25]
  Serotype 3; Post-Inj. 2 / Pre-Inj. 1 (n=94, 47) | 8.57 [6.79 to 10.8] | 1.85 [1.03 to 3.32]
  Serotype 3; Post-Inj. 2 / Pre-Inj. 2 (n=94, 47) | 2.03 [1.58 to 2.61] | 1.02 [0.701 to 1.47]
  Serotype 3; Post-Inj. 3 / Pre-Inj. 1 (n=89, 46) | 6.26 [4.82 to 8.13] | 1.24 [0.815 to 1.9]
  Serotype 3; Post-Inj. 3 / Pre-Inj. 2 (n=89, 46) | 1.46 [1.11 to 1.91] | 0.673 [0.489 to 0.925]
  Serotype 3; Post-Inj. 3 / Pre-Inj. 3 (n=88, 46) | 1.53 [1.27 to 1.86] | 0.8 [0.681 to 0.94]
  Serotype 4; Post-Inj. 1 / Pre-Inj. 1 (n=99, 48) | 17.7 [12.1 to 26.0] | 0.806 [0.665 to 0.976]
  Serotype 4; Post-Inj. 2 / Pre-Inj. 1 (n=94, 47) | 15.4 [12.3 to 19.2] | 1.27 [0.795 to 2.04]
  Serotype 4; Post-Inj. 2 / Pre-Inj. 2 (n=94, 47) | 1.84 [1.50 to 2.26] | 0.835 [0.587 to 1.19]
  Serotype 4; Post-Inj. 3 / Pre-Inj. 1 (n=89, 46) | 20.2 [15.4 to 26.3] | 1.4 [0.939 to 2.1]
  Serotype 4; Post-Inj. 3 / Pre-Inj. 2 (n=89, 46) | 2.26 [1.74 to 2.93] | 0.912 [0.606 to 1.37]
  Serotype 4; Post -nj. 3 / Pre-Inj. 3 (n=87, 46) | 1.68 [1.38 to 2.05] | 0.723 [0.564 to 0.927]

8. Primary Outcome: Geometric Mean Titers (GMTs) Against Each Serotype With the Parental of Dengue Virus Strains Before and After Vaccinations With Either CYD Dengue Vaccine or a Placebo
Description: Geometric mean titers were assessed using the Dengue Plaque Reduction Neutralization Test (PRNT).
Time Frame: Before and 28 days after each injection
Population: Geometric mean titers were assessed in the Full Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilutions)
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 99 | 49
Titers (1/dilutions)
  Serotype 1; Pre-Injection 1 (n=99, 49) | 41.4 [27.7 to 62.1] | 47.2 [26.9 to 82.7]
  Serotype 1; Post-Injection 1 (n=99, 49) | 256 [151 to 433] | 50.7 [29.5 to 87.3]
  Serotype 1; Pre-Injection 2 (n=94, 47) | 230 [138 to 384] | 86 [43.8 to 169]
  Serotype 1; Post-Injection 2 (n=94, 47) | 436 [287 to 662] | 130 [59.7 to 283]
  Serotype 1; Pre-Injection 3 (n=90, 46) | 162 [99.8 to 262] | 90.8 [46.6 to 177]
  Serotype 1; Post-Injection 3 (n=89, 46) | 267 [181 to 394] | 79.2 [42.4 to 148]
  Serotype 2; Pre-Injection 1 (n=99, 49) | 67.0 [44.0 to 102] | 68.3 [36.3 to 129]
  Serotype 2; Post-Injection 1 (n=99, 49) | 352 [210 to 592] | 62.8 [33.9 to 116]
  Serotype 2; Pre-Injection 2 (n=94, 47) | 287 [173 to 475] | 117 [57.6 to 238]
  Serotype 2; Post-Injection 2 (n=94, 47) | 647 [449 to 932] | 137 [61.4 to 306]
  Serotype 2; Pre-Injection 3 (n=90, 46) | 360 [219 to 592] | 131 [65.7 to 262]
  Serotype 2; Post-Injection 3 (n=89, 46) | 544 [378 to 782] | 132 [67 to 259]
  Serotype 3; Pre-Injection 1 (n=99, 49) | 81.9 [49.3 to 136] | 94.7 [43.6 to 206]
  Serotype 3; Post-Injection 1 (n=99, 49) | 690 [423 to 1125] | 110 [50.3 to 242]
  Serotype 3; Pre-Injection 2 (n=94, 47) | 471 [282 to 787] | 184 [80.3 to 424]
  Serotype 3; Post-Injection 2 (n=94, 47) | 1031 [704 to 1512] | 227 [92.8 to 556]
  Serotype 3; Pre-Injection 3 (n=89, 46) | 481 [300 to 772] | 144 [65.8 to 316]
  Serotype 3; Post-Injection 3 (n=89, 46) | 741 [516 to 1062] | 140 [66 to 298]
  Serotype 4; Pre-Injection 1 (n=99, 49) | 15.0 [11.6 to 19.4] | 17.5 [11.9 to 25.8]
  Serotype 4; Post-Injection 1 (n=99, 48) | 383 [262 to 559] | 19.2 [13.3 to 27.7]
  Serotype 4; Pre-Injection 2 (n=94, 47) | 178 [134 to 238] | 27.8 [16.9 to 45.8]
  Serotype 4; Post-Injection 2 (n=94, 47) | 346 [281 to 425] | 31.2 [18.1 to 53.7]
  Serotype 4; Pre-Injection 3 (n=88, 46) | 258 [192 to 347] | 37.4 [22.6 to 62.1]
  Serotype 4; Post-Injection 3 (n=89, 46) | 432 [335 to 556] | 33.4 [21.5 to 51.9]

9. Primary Outcome: Geometric Mean Titers (GMTs) of Flavivirus Immune Subjects Against Each Serotype With the Parental of Dengue Virus Strains Before and After Vaccinations With Either CYD Dengue Vaccine or a Placebo
Description: Geometric mean titers were assessed using the Dengue Plaque Reduction Neutralization Test (PRNT). Flavivirus immune subjects at baseline are defined as those subjects with ≥10 (1/dil) for at least 1 serotype with the parental dengue virus strain or for the yellow fever titer.
Time Frame: Before and 28 days after each injection
Population: Geometric mean titers were assessed in the Full Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilutions)
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 80 | 41
Titers (1/dilutions)
  Serotype 1; Pre-Injection 1 (n=80, 41) | 68.5 [44.5 to 105] | 73.1 [40.9 to 131]
  Serotype 1; Post-Injection 1 (n=80, 41) | 549 [328 to 918] | 79.8 [46.1 to 138]
  Serotype 1; Pre-Injection 2 (n=78, 39) | 430 [261 to 709] | 154 [78.5 to 303]
  Serotype 1; Post-Injection 2 (n=78, 39) | 661 [442 to 987] | 253 [116 to 553]
  Serotype 1; Pre-Injection 3 (n=74, 38) | 268 [164 to 435] | 143 [73.7 to 278]
  Serotype 1; Post-Injection 3 (n=73, 38) | 381 [256 to 566] | 126 [67.6 to 236]
  Serotype 2; Pre-Injection 1 (n=80, 41) | 124 [81.9 to 188] | 114 [59.7 to 217]
  Serotype 2; Post-Injection 1 (n=80, 41) | 816 [517 to 1290] | 103 [54.8 to 193]
  Serotype 2; Pre-Injection 2 (n=78, 39) | 591 [376 to 928] | 224 [112 to 446]
  Serotype 2; Post-Injection 2 (n=78, 39) | 978 [697 to 1374] | 271 [120 to 610]
  Serotype 2; Pre-Injection 3 (n=74, 38) | 648 [400 to 1048] | 240 [122 to 471]
  Serotype 2; Post-Injection 3 (n=73, 38) | 835 [584 to 1193] | 242 [126 to 463]
  Serotype 3; Pre-Injection 1 (n=80, 41) | 159 [93.5 to 271] | 168 [74.3 to 380]
  Serotype 3; Post-Injection 1 (n=80, 41) | 1263 [764 to 2088] | 202 [89.3 to 455]
  Serotype 3; Pre-Injection 2 (n=78, 39) | 879 [531 to 1455] | 387 [170 to 878]
  Serotype 3; Post-Injection 2 (n=78, 39) | 1426 [950 to 2141] | 497 [204 to 1210]
  Serotype 3; Pre-Injection 3 (n=74, 38) | 776 [481 to 1251] | 272 [122 to 606]
  Serotype 3; Post-Injection 3 (n=73, 38) | 1031 [700 to 1519] | 266 [125 to 566]
  Serotype 4; Pre-Injection 1 (n=80, 41) | 19.5 [14.6 to 26.1] | 22.4 [14.6 to 34.3]
  Serotype 4; Post-Injection 1 (n=80, 40) | 467 [325 to 672] | 25.2 [17.1 to 37.1]
  Serotype 4; Pre-Injection 2 (n=78, 39) | 220 [164 to 295] | 39.5 [23.1 to 67.6]
  Serotype 4; Post-Injection 2 (n=78, 39) | 377 [303 to 470] | 45.3 [25.1 to 81.8]
  Serotype 4; Pre-Injection 3 (n=73, 38) | 313 [231 to 424] | 53.9 [31.7 to 91.8]
  Serotype 4; Post-Injection 3 (n=73, 38) | 485 [374 to 628] | 46.5 [29.3 to 73.6]

10. Primary Outcome: Geometric Mean Titer Ratios (GMTRs) of Flavivirus naïve Subjects Against Each Serotype With the Parental of Dengue Virus Strains Before and After Vaccinations With Either CYD Dengue Vaccine or a Placebo
Description: Geometric mean titers were assessed using the Dengue Plaque Reduction Neutralization Test (PRNT). Flavivirus naïve subjects at baseline are defined as those subjects with <10 (1/dil) for all serotypes with parental dengue virus strains and for yellow fever titer.
Time Frame: Before and 28 days after each injection
Population: Geometric mean titer ratios were assessed in the Full Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer ratio
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 19 | 8
Titer ratio
  Serotype 1; Post-Inj. 1 / Pre-Inj. 1 (n=19, 8) | 1.03 [0.639 to 1.67] | 0.5 [0.5 to 0.5]
  Serotype 1; Post-Inj. 2 / Pre-Inj. 1 (n=16, 8) | 5.73 [1.89 to 17.3] | 0.5 [0.5 to 0.5]
  Serotype 1; Post-Inj. 2 / Pre-Inj. 2 (n=16, 8) | 3.25 [1.18 to 8.93] | 0.5 [0.5 to 0.5]
  Serotype 1; Post-Inj. 3 / Pre-Inj. 1 (n=16, 8) | 5.34 [2.25 to 12.7] | 0.861 [0.238 to 3.11]
  Serotype 1; Post-Inj. 3 / Pre-Inj. 2 (n=16, 8) | 3.03 [1.35 to 6.80] | 0.861 [0.238 to 3.11]
  Serotype 1; Post-Inj. 3 / Pre-Inj. 3 (n=16, 8) | 2.19 [1.37 to 3.48] | 0.446 [0.342 to 0.584]
  Serotype 2; Post-Inj. 1 / Pre-Inj. 1 (n=19, 8) | 1.02 [0.527 to 1.99] | 0.5 [0.5 to 0.5]
  Serotype 2; Post-Inj. 2 / Pre-Inj. 1 (n=16, 8) | 8.62 [3.49 to 21.3] | 0.5 [0.5 to 0.5]
  Serotype 2; Post-Inj. 2 / Pre-Inj. 2 (n=16, 8) | 6.02 [2.37 to 15.3] | 0.5 [0.5 to 0.5]
  Serotype 2; Post-Inj. 3 / Pre-Inj. 1 (n=16, 8) | 7.67 [4.19 to 14.0] | 0.737 [0.294 to 1.85]
  Serotype 2; Post-Inj. 3 / Pre-Inj. 2 (n=16, 8) | 5.36 [2.73 to 10.5] | 0.737 [0.294 to 1.85]
  Serotype 2; Post -nj. 3 / Pre-Inj. 3 (n=16, 8) | 2.37 [1.35 to 4.17] | 0.538 [0.453 to 0.639]
  Serotype 3; Post-Inj. 1 / Pre-Inj. 1 (n=19, 8) | 5.41 [2.80 to 10.5] | 0.5 [0.5 to 0.5]
  Serotype 3; Post-Inj. 2 / Pre-Inj. 1 (n=16, 8) | 21.2 [10.5 to 42.9] | 0.5 [0.5 to 0.5]
  Serotype 3; Post-Inj. 2 / Pre-Inj. 2 (n=16, 8) | 7.58 [3.12 to 18.4] | 0.5 [0.5 to 0.5]
  Serotype 3; Post-Inj. 3 / Pre-Inj. 1 (n=16, 8) | 16.3 [9.65 to 27.7] | 0.678 [0.33 to 1.39]
  Serotype 3; Post-Inj. 3 / Pre-Inj. 2 (n=16, 8) | 5.83 [3.17 to 10.7] | 0.678 [0.33 to 1.39]
  Serotype 3; Post-Inj. 3 / Pre-Inj. 3 (n=15, 8) | 3.35 [1.92 to 5.84] | 0.524 [0.469 to 0.587]
  Serotype 4; Post-Inj. 1 / Pre-Inj. 1 (n=19, 8) | 16.5 [4.58 to 59.1] | 0.5 [0.5 to 0.5]
  Serotype 4; Post-Inj. 2 / Pre-Inj. 1 (n=16, 8) | 22.7 [12.8 to 40.3] | 0.5 [0.5 to 0.5]
  Serotype 4; Post-Inj. 2 / Pre-Inj. 2 (n=16, 8) | 3.15 [1.63 to 6.09] | 0.5 [0.5 to 0.5]
  Serotype 4; Post-Inj. 3 / Pre-Inj. 1 (n=16, 8) | 25.5 [11.6 to 55.9] | 0.701 [0.414 to 1.19]
  Serotype 4; Post-Inj. 3 / Pre-Inj. 2 (n=16, 8) | 3.53 [1.71 to 7.26] | 0.701 [0.414 to 1.19]
  Serotype 4; Post-Inj. 3 / Pre-Inj. 3 (n=15, 8) | 2.55 [1.37 to 4.75] | 0.578 [0.401 to 0.832]

11. Primary Outcome: Percentage of Participants Reporting Solicited Injection-Site and Systemic Reactions Following Any and Each Vaccination With Either CYD Dengue Vaccine or a Placebo
Description: Injection-site reactions: Pain, Erythema, and Swelling. Systemic reactions: Fever, Headache, Malaise, Myalgia, and Asthenia. Grade 3 Injection-site reactions (9 to 11 years): Pain, Incapacitating, unable to perform usual activities; Erythema and Swelling, ≥5 cm. Grade 3 Injection site reactions (≥12 years): Pain, Significant; prevents daily activity; Erythema and Swelling, >10 cm. Grade 3 Systemic reactions: Fever, ≥39˚C; Headache, Malaise, Myalgia, and Asthenia, Significant; prevents daily activity.
Time Frame: Day 0 up to Day 14 post each vaccination
Population: Solicited injection-site and systemic reactions were assessed in the Safety Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 100 | 50
Percentage of participants
  Injection-site Pain; Post-Any Injection (N=100,49) | 40 | 40.8
  Grade 3 Inj.-site Pain; Post-Any Inj. (N=100,49) | 0 | 4.1
  Inj.-site Erythema; Post-Any Inj. (N=100,49) | 4.0 | 2
  Gr 3 Inj.-site Erythema; Post-Any Inj. (N=100,49) | 0 | 0
  Inj.-site Swelling; Post-Any Inj. (N=100,49) | 5.0 | 4.1
  Gr 3 Inj.-site Swelling; Post-Any Inj. (N=100,49) | 0 | 0
  Injection-site Pain; Post-Injection 1 (N=99,49) | 26.3 | 30.6
  Gr 3 Inj.-site Pain; Post-Inj. 1 (N=99,49) | 0 | 2
  Inj.-site Erythema; Post-Inj. 1 (N=99,49) | 1.0 | 2
  Gr 3 Inj.-site Erythema; Post-Inj. 1 (N=99,49) | 0 | 0
  Inj.-site Swelling; Post-Inj. 1 (N=99,49) | 2.0 | 4.1
  Gr 3 Inj.-site Swelling; Post-Inj. 1 (N=99,49) | 0 | 0
  Injection-site Pain; Post-Injection 2 (N=93,47) | 21.5 | 14.9
  Gr 3 Inj.-site Pain; Post-Inj. 2 (N=93,47) | 0 | 2.1
  Inj.-site Erythema; Post-Inj. 2 (N=93,47) | 3.2 | 0
  Gr 3 Inj.-site Erythema; Post-Inj. 2 (N=93,47) | 0 | 0
  Inj.-site Swelling; Post-Inj. 2 (N=93,47) | 2.2 | 0
  Gr 3 Inj.-site Swelling; Post-Inj. 2 (N=93,47) | 0 | 0
  Injection-site Pain; Post-Injection 3 (N=89,45) | 16.9 | 15.6
  Gr 3 Inj.-site Pain; Post-Inj. 3 (N=89,45) | 0 | 2.2
  Inj.-site Erythema; Post-Inj. 3 (N=89,45) | 0 | 0
  Gr 3 Inj.-site Erythema; Post-Inj. 3 (N=89,45) | 0 | 0
  Inj.-site Swelling; Post-Inj. 3 (N=89,45) | 1.1 | 0
  Gr 3 Inj.-site Swelling; Post-Inj. 3 (N=89,45) | 0 | 0
  Fever; Post-Any Injection (N=100, 49) | 30.0 | 18.4
  Grade 3 Fever; Post-Any Injection (N=100, 49) | 8.0 | 6.1
  Headache; Post-Any Injection (N=100, 49) | 61.0 | 51
  Grade 3 Headache; Post-Any Injection (N=100, 49) | 15.0 | 20.4
  Malaise; Post-Any Injection (N=100, 49) | 40.0 | 32.7
  Grade 3 Malaise; Post-Any Injection (N=100, 49) | 11.0 | 6.1
  Myalgia; Post-Any Injection (N=100, 49) | 42.0 | 42.9
  Grade 3 Myalgia; Post-Any Injection (N=100, 49) | 6.0 | 8.2
  Asthenia; Post-Any Injection (N=100, 49) | 35.0 | 20.4
  Grade 3 Asthenia; Post-Any Injection (N=100, 49) | 8.0 | 4.1
  Fever; Post-Injection 1 (N=98, 48) | 15.3 | 10.4
  Grade 3 Fever; Post-Injection 1 (N=98, 48) | 3.1 | 2.1
  Headache; Post-Injection 1 (N=99, 49) | 48.5 | 40.8
  Grade 3 Headache; Post-Injection 1 (N=99, 49) | 8.1 | 10.2
  Malaise; Post-Injection 1 (N=99, 49) | 31.3 | 18.4
  Grade 3 Malaise; Post-Injection 1 (N=99, 49) | 3.0 | 2
  Myalgia; Post-Injection 1 (N=99, 49) | 32.3 | 30.6
  Grade 3 Myalgia; Post-Injection 1 (N=99, 49) | 2.0 | 6.1
  Asthenia; Post-Injection 1 (N=99, 49) | 22.2 | 10.2
  Grade 3 Asthenia; Post-Injection 1 (N=99, 49) | 4.0 | 4.1
  Fever; Post-Injection 2 (N=92, 47) | 8.7 | 4.3
  Grade 3 Fever; Post-Injection 2 (N=92, 47) | 2.2 | 0
  Headache; Post-Injection 2 (N=94, 47) | 28.7 | 34
  Grade 3 Headache; Post-Injection 2 (N=94, 47) | 5.3 | 6.4
  Malaise; Post-Injection 2 (N=94, 47) | 18.1 | 17
  Grade 3 Malaise; Post-Injection 2 (N=94, 47) | 6.4 | 4.3
  Myalgia; Post-Injection 2 (N=94, 47) | 20.2 | 21.3
  Grade 3 Myalgia; Post-Injection 2 (N=94, 47) | 3.2 | 4.3
  Asthenia; Post-Injection 2 (N=94, 47) | 12.8 | 14.9
  Grade 3 Asthenia; Post-Injection 2 (N=94, 47) | 3.2 | 0
  Fever; Post-Injection 3 (N=82, 43) | 11.0 | 7
  Grade 3 Fever; Post-Injection 3 (N=82, 43) | 3.7 | 7
  Headache; Post-Injection 3 (N=89, 45) | 27.0 | 20
  Grade 3 Headache; Post-Injection 3 (N=89, 45) | 5.6 | 8.9
  Malaise; Post-Injection 3 (N=89, 45) | 15.7 | 11.1
  Grade 3 Malaise; Post-Injection 3 (N=89, 45) | 2.2 | 0
  Myalgia; Post-Injection 3 (N=89, 45) | 20.2 | 11.1
  Grade 3 Myalgia; Post-Injection 3 (N=89, 45) | 2.2 | 0
  Asthenia; Post-Injection 3 (N=89, 45) | 14.6 | 4.4
  Grade 3 Asthenia; Post-Injection 3 (N=89, 45) | 2.2 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Day 0 (post-vaccination) up to Day 14 post-Injection 3
Arm/Group | CYD Dengue Vaccine Group | Control Group
Serious Adverse Events (participants affected / at risk) | 5/100 | 3/50
Other Adverse Events (participants affected / at risk) | 61/100 | 25/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYD Dengue Vaccine Group (N=100) | Control Group (N=50)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intra uterine death (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | CYD Dengue Vaccine Group (N=100) | Control Group (N=50)
Limb injury (Injury, poisoning and procedural complications) | 6 (6) | 4 (4)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 4 (4)
Lymphadenopathy (Blood and lymphatic system disorders) | 9 (9) | 1 (2)
Headache: Post Any Injection (Nervous system disorders) | 61 (61) | 25/49 (25)
Conjunctivitis (Eye disorders) | 11 (11) | 7 (7)
Injection site Pain; Post Any Injection (General disorders) | 40 (40) | 20/49 (20)
Injection site Swelling; Post Any Injection (General disorders) | 5 (5) | 2/49 (2)
Fever; Post Any Injection (General disorders) | 30 (30) | 9/49 (9)
Malaise; Post-Any Injection (General disorders) | 40 (40) | 16/49 (16)
Asthenia; Post-Any Injection (General disorders) | 35 (35) | 10/49 (10)
Abdominal pain (Gastrointestinal disorders) | 12 (16) | 4 (6)
Nausea (Gastrointestinal disorders) | 8 (11) | 0 (0)
Vomiting (Gastrointestinal disorders) | 7 (7) | 2 (2)
Myalgia; Post-Any Injection (Musculoskeletal and connective tissue disorders) | 42 (42) | 21/49 (21)
Nasopharyngitis (Infections and infestations) | 12 (12) | 6 (6)
Rhinitis (Infections and infestations) | 6 (7) | 2 (2)
Tonsillitis (Infections and infestations) | 5 (5) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 18 (19) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications